CLINICAL TRIAL: NCT02647775
Title: Hemodynamic and Inflammatory Responses in Thoracic Surgery: Hemodynamic and Inflammatory Responses Following Video-assisted Thoracoscopic Surgery
Brief Title: Hemodynamic and Inflammatory Responses in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-IRB-104-7159A3
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Video-Assisted Thoracic Surgery
Keywords: Thoracoscopic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multi-port VATS (Other): Multi-port VATS is an operative method
  Interventions: Procedure: multi-port VATS
- single-port VATS (Other): Single-port VATS is an operative method
  Interventions: Procedure: single-port VATS

INTERVENTIONS:
Procedure: multi-port VATS — Patients with thoracic surgical diseases who underwent VATS will be recruited into this study to investigate the postoperative pain , physiologic and immunologic impacts of two different approaches for minimally invasive thoracic surgery.
  Arms: multi-port VATS
Procedure: single-port VATS — Patients with thoracic surgical diseases who underwent VATS will be recruited into this study to investigate the postoperative pain , physiologic and immunologic impacts of two different approaches for minimally invasive thoracic surgery.
  Arms: single-port VATS

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) for thoracic surgery is practical, has been shown to reduce postoperative discomfort, and has improved cosmetic results when compare to open thoracotomy. The specific aims of this project are: to clarify the physiologic and immunologic effects of different approaches for minimally invasive thoracic surgery: (1) multiple-port VATS; (2) single-port VATS

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) was first reported in the early 1990s. Since then, the safety and efficacy of thoracoscopy for diagnosing and treating pleural, pulmonary, and mediastinal disease has been demonstrated with similar oncological results, which were confirmed by multiple clinical studies. Although VATS for thoracic surgery is practical, has been shown to reduce postoperative discomfort, and has improved cosmetic results when compare to open thoracotomy, unfortunately chronic thoracic wound discomfort and postoperative neuralgia were found in a significant portion of patients .

Recently, a minimally invasive approach that is different from the conventional multiport thoracoscopic technique is gradually becoming of great interest in the diagnosis and treatment of thoracic surgical disease. Single-port VATS is one of the most promising emerging surgical techniques which allows the surgeon to perform a majority of thoracic surgeries and with similar perioperative outcomes that are comparable with the conventional multiport technique. However, a very limited number of clinical studies have demonstrated the advantages of single port VATS in postoperative pain reduction, when comparing to the traditional multiport thoracoscopic approach.

To clarify the physiologic and immunologic effects of different approaches for minimally invasive thoracic surgery, investigators aim to compare the perioperative physiological changes, immunological responses, and postoperative pain between standard (multi-port) transthoracic thoracoscopic and single-port transthoracic thoracoscopic surgery for thoracic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with thoracic surgical diseases(lung cancer. mediastinal tumor. solitary pulmonary lesion. pneumothorax) who will be underwent video-assisted thoracic surgery

Exclusion Criteria:

* Unresectable mediastinal tumor
* Previous history of ipsilateral pulmonary resection
* Patients with complex cardiopulmonary dysfunction
* Unresectable pulmonary hilar tumor

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pain score | beginning at 3 hours after surgery until 5 days
  Numerical Rating Scale (NRS) or Wong-Baker Face Pain Rating Scale

SECONDARY OUTCOMES:
Complication | beginning at 3 hours after surgery until 30 days
  Yes/No
Mean arterial pressure | beginning 20 min before the start of surgery until 20 min after the surgery.
  MAP; mmHg
Heart rate | beginning 20 min before the start of surgery until 20 min after the surgery.
  HR; beats per min [bpm]
Cardiac index | beginning 20 min before the start of surgery until 20 min after the surgery.
  CI; L/[min·m2]
Systemic vascular resistance index | beginning 20 min before the start of surgery until 20 min after the surgery.
  SVRI; [dyn·s]/[cm-5·m2]
Global end-diastolic volume index | beginning 20 min before the start of surgery until 20 min after the surgery.
  GEDVI; mL/m2
Leukocyte subset analysis | preoperation till 5 days after surgery
  10^3/ul
Intracellular oxidative activity of neutrophils | preoperation till 5 days after surgery
  ratio compared with preoperation
Inducible nitric oxide synthase expression in monocytes | preoperation till 5 days after surgery
  Arbitrary intensity
Interleukin-6 | preoperation till 5 days after surgery
  pg/ml
C-reactive protein | preoperation till 5 days after surgery
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hen Liu, Principal Investigator — Chang Gung Memorial Hospital; Hung-Pin Liu, Principal Investigator — Chang Gung Memorial Hospital; Yi-Cheng Wu, Principal Investigator — Chang Gung Memorial Hospital; Ming-Ju Hsieh, Principal Investigator — Chang Gung Memorial Hospital; Wei-Hsun Chen, Principal Investigator — Chang Gung Memorial Hospital; Yen Chu, Principal Investigator — Chang Gung Memorial Hospital; Chien-Ying Liu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Nagahiro I, Andou A, Aoe M, Sano Y, Date H, Shimizu N. Pulmonary function, postoperative pain, and serum cytokine level after lobectomy: a comparison of VATS and conventional procedure. Ann Thorac Surg. 2001 Aug;72(2):362-5. doi: 10.1016/s0003-4975(01)02804-1. PMID 11515867
- [Background] Flores RM, Park BJ, Dycoco J, Aronova A, Hirth Y, Rizk NP, Bains M, Downey RJ, Rusch VW. Lobectomy by video-assisted thoracic surgery (VATS) versus thoracotomy for lung cancer. J Thorac Cardiovasc Surg. 2009 Jul;138(1):11-8. doi: 10.1016/j.jtcvs.2009.03.030. PMID 19577048
- [Background] Onaitis MW, Petersen RP, Balderson SS, Toloza E, Burfeind WR, Harpole DH Jr, D'Amico TA. Thoracoscopic lobectomy is a safe and versatile procedure: experience with 500 consecutive patients. Ann Surg. 2006 Sep;244(3):420-5. doi: 10.1097/01.sla.0000234892.79056.63. PMID 16926568
- [Background] Sihoe AD, Au SS, Cheung ML, Chow IK, Chu KM, Law CY, Wan M, Yim AP. Incidence of chest wall paresthesia after video-assisted thoracic surgery for primary spontaneous pneumothorax. Eur J Cardiothorac Surg. 2004 Jun;25(6):1054-8. doi: 10.1016/j.ejcts.2004.02.018. PMID 15145009
- [Background] Rocco G, Martin-Ucar A, Passera E. Uniportal VATS wedge pulmonary resections. Ann Thorac Surg. 2004 Feb;77(2):726-8. doi: 10.1016/S0003-4975(03)01219-0. PMID 14759479
- [Background] Gonzalez-Rivas D, Fieira E, Mendez L, Garcia J. Single-port video-assisted thoracoscopic anatomic segmentectomy and right upper lobectomy. Eur J Cardiothorac Surg. 2012 Dec;42(6):e169-71. doi: 10.1093/ejcts/ezs482. Epub 2012 Aug 24. PMID 22922693
- [Background] Gonzalez-Rivas D, de la Torre M, Fernandez R, Garcia J. Video: Single-incision video-assisted thoracoscopic right pneumonectomy. Surg Endosc. 2012 Jul;26(7):2078-9. doi: 10.1007/s00464-011-2127-x. Epub 2012 Jan 11. PMID 22234590
- [Background] Gonzalez-Rivas D, Fieira E, Delgado M, de la Torre M, Mendez L, Fernandez R. Uniportal video-assisted thoracoscopic sleeve lobectomy and other complex resections. J Thorac Dis. 2014 Oct;6(Suppl 6):S674-81. doi: 10.3978/j.issn.2072-1439.2014.09.17. PMID 25379210
- [Background] Wang BY, Liu CY, Hsu PK, Shih CS, Liu CC. Single-incision versus multiple-incision thoracoscopic lobectomy and segmentectomy: a propensity-matched analysis. Ann Surg. 2015 Apr;261(4):793-9. doi: 10.1097/SLA.0000000000000712. PMID 24836148
- [Background] Ocakcioglu I, Alpay L, Demir M, Kiral H, Akyil M, Dogruyol T, Tezel C, Baysungur V, Yalcinkaya I. Is single port enough in minimally surgery for pneumothorax? Surg Endosc. 2016 Jan;30(1):59-64. doi: 10.1007/s00464-015-4161-6. Epub 2015 Mar 24. PMID 25801108
- [Background] Swanstrom LL, Kurian A, Dunst CM, Sharata A, Bhayani N, Rieder E. Long-term outcomes of an endoscopic myotomy for achalasia: the POEM procedure. Ann Surg. 2012 Oct;256(4):659-67. doi: 10.1097/SLA.0b013e31826b5212. PMID 22982946
- [Background] Ujiki MB, Yetasook AK, Zapf M, Linn JG, Carbray JM, Denham W. Peroral endoscopic myotomy: A short-term comparison with the standard laparoscopic approach. Surgery. 2013 Oct;154(4):893-7; discussion 897-900. doi: 10.1016/j.surg.2013.04.042. PMID 24074429
- [Background] Liu YH, Chu Y, Wu YC, Yeh CJ, Liu CY, Hsieh MJ, Yuan HC, Ko PJ, Liu HP. Natural orifice surgery in thoracic surgery. J Thorac Dis. 2014 Jan;6(1):61-3. doi: 10.3978/j.issn.2072-1439.2014.01.02. No abstract available. PMID 24455178
- [Background] Takata M, Watanabe G, Ushijima T, Ishikawa N. A novel internal thoracic artery harvesting technique via subxiphoid approach--for the least invasive coronary artery bypass grafting. Interact Cardiovasc Thorac Surg. 2009 Nov;9(5):891-2. doi: 10.1510/icvts.2009.212282. Epub 2009 Aug 31. PMID 19720658
- [Background] St Peter SD, Sharp SW, Ostlie DJ, Snyder CL, Holcomb GW 3rd, Sharp RJ. Use of a subxiphoid incision for pectus bar placement in the repair of pectus excavatum. J Pediatr Surg. 2010 Jun;45(6):1361-4. doi: 10.1016/j.jpedsurg.2010.02.115. PMID 20620345
- [Background] Taniguchi Y, Suzuki Y, Suda T, Inoue T, Araki K, Ito N, Okada K, Ishiguro K, Nakamura H, Ohgi S. Video-assisted thoracoscopic bilateral lung metastasectomy with a subxiphoid access port. J Thorac Cardiovasc Surg. 2005 Sep;130(3):916-7. doi: 10.1016/j.jtcvs.2005.03.039. No abstract available. PMID 16153963
- [Background] Suda T, Ashikari S, Tochii S, Sugimura H, Hattori Y. Single-incision subxiphoid approach for bilateral metastasectomy. Ann Thorac Surg. 2014 Feb;97(2):718-9. doi: 10.1016/j.athoracsur.2013.06.123. PMID 24484826
- [Background] Liu CC, Wang BY, Shih CS, Liu YH. Subxiphoid single-incision thoracoscopic left upper lobectomy. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3250-1. doi: 10.1016/j.jtcvs.2014.08.033. Epub 2014 Aug 23. No abstract available. PMID 25240526
- [Background] Craig SR, Leaver HA, Yap PL, Pugh GC, Walker WS. Acute phase responses following minimal access and conventional thoracic surgery. Eur J Cardiothorac Surg. 2001 Sep;20(3):455-63. doi: 10.1016/s1010-7940(01)00841-7. PMID 11509263
- [Background] Martins PS, Kallas EG, Neto MC, Dalboni MA, Blecher S, Salomao R. Upregulation of reactive oxygen species generation and phagocytosis, and increased apoptosis in human neutrophils during severe sepsis and septic shock. Shock. 2003 Sep;20(3):208-12. doi: 10.1097/01.shk.0000079425.52617.db. PMID 12923490
- [Background] Haugen TS, Skjonsberg OH, Kahler H, Lyberg T. Production of oxidants in alveolar macrophages and blood leukocytes. Eur Respir J. 1999 Nov;14(5):1100-5. doi: 10.1183/09031936.99.14511009. PMID 10596697
- [Background] Romeo C, Impellizzeri P, Antonuccio P, Turiaco N, Cifala S, Gentile C, Passaniti M, Marini H, Squadrito F, Altavilla D. Peritoneal macrophage activity after laparoscopy or laparotomy. J Pediatr Surg. 2003 Jan;38(1):97-101; discussion 97-101. doi: 10.1053/jpsu.2003.50019. PMID 12592628
- [Background] Ni Choileain N, Redmond HP. Cell response to surgery. Arch Surg. 2006 Nov;141(11):1132-40. doi: 10.1001/archsurg.141.11.1132. PMID 17116807
- [Background] Wichmann MW, Huttl TP, Winter H, Spelsberg F, Angele MK, Heiss MM, Jauch KW. Immunological effects of laparoscopic vs open colorectal surgery: a prospective clinical study. Arch Surg. 2005 Jul;140(7):692-7. doi: 10.1001/archsurg.140.7.692. PMID 16027336
- [Background] Ordemann J, Jacobi CA, Schwenk W, Stosslein R, Muller JM. Cellular and humoral inflammatory response after laparoscopic and conventional colorectal resections. Surg Endosc. 2001 Jun;15(6):600-8. doi: 10.1007/s004640090032. Epub 2001 Apr 3. PMID 11591950
- [Background] Ng CS, Wan S, Hui CW, Lee TW, Underwood MJ, Yim AP. Video-assisted thoracic surgery for early stage lung cancer - can short-term immunological advantages improve long-term survival? Ann Thorac Cardiovasc Surg. 2006 Oct;12(5):308-12. PMID 17095971
- [Background] Ng CS, Whelan RL, Lacy AM, Yim AP. Is minimal access surgery for cancer associated with immunologic benefits? World J Surg. 2005 Aug;29(8):975-81. doi: 10.1007/s00268-005-0029-6. PMID 15981046
- [Background] Natsume T, Kawahira H, Hayashi H, Nabeya Y, Akai T, Horibe D, Shuto K, Akutsu Y, Matsushita K, Nomura F, Matsubara H. Low peritoneal and systemic inflammatory response after laparoscopy-assisted gastrectomy compared to open gastrectomy. Hepatogastroenterology. 2011 Mar-Apr;58(106):659-62. PMID 21661448
- [Background] von Delius S, Wilhelm D, Feussner H, Sager J, Becker V, Schuster T, Schneider A, Schmid RM, Meining A. Natural orifice transluminal endoscopic surgery: cardiopulmonary safety of transesophageal mediastinoscopy. Endoscopy. 2010 May;42(5):405-12. doi: 10.1055/s-0029-1243948. Epub 2010 Mar 4. PMID 20205072
- [Background] von Delius S, Schorn A, Grimm M, Schneider A, Wilhelm D, Schuster T, Stangassinger M, Feussner H, Schmid RM, Meining A. Natural-orifice transluminal endoscopic surgery: low-pressure pneumoperitoneum is sufficient and is associated with an improved cardiopulmonary response (PressurePig Study). Endoscopy. 2011 Sep;43(9):808-15. doi: 10.1055/s-0030-1256559. Epub 2011 Jul 5. PMID 21732271
- [Background] Navarro-Ripoll R, Martinez-Palli G, Guarner-Argente C, Cordova H, Martinez-Zamora MA, Comas J, Rodriguez de Miguel C, Beltran M, Rodriguez-D'Jesus A, Hernandez-Cera C, Llach J, Balust J, Fernandez-Esparrach G. On-demand endoscopic CO2 insufflation with feedback pressure regulation during natural orifice transluminal endoscopic surgery (NOTES) peritoneoscopy induces minimal hemodynamic and respiratory changes. Gastrointest Endosc. 2012 Aug;76(2):388-95. doi: 10.1016/j.gie.2011.10.015. PMID 22817790
- [Background] Chu Y, Liu CY, Wu YC, Hsieh MJ, Chen TP, Chao YK, Wu CY, Yuan HC, Ko PJ, Liu YH, Liu HP. Comparison of hemodynamic and inflammatory changes between transoral and transthoracic thoracoscopic surgery. PLoS One. 2013;8(1):e50338. doi: 10.1371/journal.pone.0050338. Epub 2013 Jan 3. PMID 23300944
- [Background] Lu HY, Chu Y, Wu YC, Liu CY, Hsieh MJ, Chao YK, Wu CY, Yuan HC, Ko PJ, Liu YH, Liu HP. Hemodynamic and inflammatory responses following transumbilical and transthoracic lung wedge resection in a live canine model. Int J Surg. 2015 Apr;16(Pt A):116-122. doi: 10.1016/j.ijsu.2015.02.027. Epub 2015 Mar 11. PMID 25769396